CLINICAL TRIAL: NCT06346561
Title: The Efficacy of Dexmedetomidine Versus Labetalol In Providing Controlled Hypotension In Dacryocystorhinostomy SurgeryA Comparative Randomized Prospective Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Aboesoud Mahmoud, Resident of Anesthesia, Intensive Care and Pain management Sohag university hospital., Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-24-02-10MS
Record Dates: First submitted 2024-03-10; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Nasolacrimal Duct Obstruction
MeSH Terms: conditions — Lacrimal Duct Obstruction | interventions — Dexmedetomidine; Labetalol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Active Comparator)
  Interventions: Drug: Dexmedetomidine; Drug: Labetalol
- Labetalol group (Active Comparator)
  Interventions: Drug: Dexmedetomidine; Drug: Labetalol

INTERVENTIONS:
Drug: Dexmedetomidine — the reduction of controlled hypotension and the control of hemodynamic responses of the body
Drug: Labetalol — the reduction of controlled hypotension and the control of hemodynamic responses of the body

SUMMARY:
The most important symptoms of nasolacrimal duct obstruction are excessive tearing and mucoid discharge.

The proposed treatment in this regard is dacryocystorhinostomy (DCR) surgery. Therefore, hemostasis is of great significance in performing DCR surgery. In this regard, the reduction of controlled hypotension and the control of hemodynamic responses of the body to stress effectively reduce the bleeding volume during surgery.

Hence, there is no enough studies about controlled hypotension in DCR we decided to perform such a comparison between the effect of dexmedetomidine and labetalol in providing controlled hypotension during DCR surgery.

ELIGIBILITY:
Inclusion Criteria:

* physical status I or II according to ASA classification, age between ( 18 - 60 years )

Exclusion Criteria:

* Patients with physical status other than 1 and 2 according to ASA classification as :Hypertension, Diabetes mellitus, Ischemic heart diseases, Severe anemia, COPD, History of stroke, Impaired liver or renal function, Increase intercranial tension.
* Allergy to any of the drug included in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Assess non invasive blood pressure during DCR surgery To compare between the effect of dexmedetomidine and labetalol in providing controlled hypotension. | 5 months
  Controlled Hypotension In Dacryocystorhinostomy Surgery By:
  Dexmedetomidine is a potent α2 adrenergic agonist. Labetalol is a beta-adrenergic blocker agent with alpha1 and beta-adrenergic receptors blocking action

SECONDARY OUTCOMES:
Effectiveness of dexamedetomidine for prolongation of postoperative analgesia. | 5 months
  Dexmedetomidine is a potent α2 adrenergic agonist. One of the highest densities of α2 receptors is located in the pontine locus cereleus, an important nucleus mediating sympathetic nervous system function. It has sedative, anxiolytic, hypnotic, analgesic, and sympatholytic properties.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vinciguerra A, Nonis A, Resti AG, Bussi M, Trimarchi M. Impact of Post-Surgical Therapies on Endoscopic and External Dacryocystorhinostomy: Systematic Review and Meta-Analysis. Am J Rhinol Allergy. 2020 Nov;34(6):846-856. doi: 10.1177/1945892420945218. Epub 2020 Jul 23. PMID 32703027
- [Background] Heindl LM, Junemann AG, Kruse FE, Holbach LM. Tumors of the lacrimal drainage system. Orbit. 2010 Oct;29(5):298-306. doi: 10.3109/01676830.2010.492887. PMID 20958177
- [Background] Degoute CS, Dubreuil C, Ray MJ, Guitton J, Manchon M, Banssillon V, Saumet JL. Effects of posture, hypotension and locally applied vasoconstriction on the middle ear microcirculation in anaesthetized humans. Eur J Appl Physiol Occup Physiol. 1994;69(5):414-20. doi: 10.1007/BF00865405. PMID 7875138
- [Background] Alicandri-Ciufelli M, Pingani L, Maccarrone F, Anschuetz L, Mariano D, Galeazzi GM, Presutti L, Molinari G. Validation of the Modena bleeding score in endoscopic sinus surgery. Braz J Otorhinolaryngol. 2022 Jul-Aug;88(4):602-606. doi: 10.1016/j.bjorl.2020.08.006. Epub 2020 Sep 30. PMID 33279423
- [Background] Rahimzadeh P, Faiz SH, Alebouyeh MR. Effects of premedication with metoprolol on bleeding and induced hypotension in nasal surgery. Anesth Pain Med. 2012 Winter;1(3):157-61. doi: 10.5812/kowsar.22287523.3408. Epub 2012 Jan 1. PMID 24904785